CLINICAL TRIAL: NCT03090906
Title: Clinical and Histological Analysis of Soft Tissue Volume Gain and Stability Around Dental Implants Using Autogenous Subepithelial Connective Tissue Grafts Harvested From the Palate or Tuberosity. A Randomized Controlled Clinical Study
Brief Title: Soft Tissue Volume Gain and Stability Comparing Palate and Tuberosity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Osteology Foundation (Other)
Responsible Party: Principal Investigator, Ernest Rojo Xicart, Professor Section of Periodontology, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER- ECL-2011-10-NF
Record Dates: First submitted 2017-01-29; First posted 2017-03-27 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Tooth Loss; Recession, Gingival
Keywords: volume gain; soft tissue augmentation; dental implants; histology
MeSH Terms: conditions — Tooth Loss; Gingival Recession

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: SCTG from palate (Experimental): Soft tissue augmentation palate
  Interventions: Procedure: Soft tissue augmentation palate; Device: Intraoral optical scan
- Test group: SCTG from tuberosity (Experimental): Soft tissue augmentation tuberosity
  Interventions: Procedure: Soft tissue augmentation tuberosity; Device: Intraoral optical scan

INTERVENTIONS:
Procedure: Soft tissue augmentation palate — Recipient site: Intrasulcular incision at the buccal side of the implant extending in one adjacent tooth for each side and a partial-thickness mucosal ﬂap raised. The connective tissue was secured with suture. Allocation to either treatment was performed according to a randomization table.
  Donor site A double-bladed scalpel handle 1,5mm was used in both areas to obtain the same thickness.
  Palate (CG) The double incision was made approximately 2 to 3 mm apical to the gingival margins of premolars. The donor tissue was removed and cross-mattress sutures were used to approximate the wound on the palate.
  In both groups the epithelial collar removed. Graft required dimensions for both groups:10mm height, 12mm length and 1,5mm thick.
  Other Names: subepithelial connective tissue graft
  Arms: Control group: SCTG from palate
Procedure: Soft tissue augmentation tuberosity — Recipient site: Intrasulcular incision at the buccal side of the implant extending in one adjacent tooth for each side and a partial-thickness mucosal ﬂap raised. The connective tissue was secured with suture. Allocation to either treatment was performed according to a randomization table.
  Donor site A double-bladed scalpel handle 1,5mm was used in both areas to obtain the same thickness.
  Tuberosity (TG) The double incision was made from the distal of the terminal tooth. A second incision was made perpendicular to the linear incision at a distal point, which joined the two linear incisions. The graft was removed and a crossed horizontal suspension suture was used.
  Epithelial collar removed. Graft required dimensions for both groups:10mm height, 12mm length and 1,5mm thick.
  Other Names: subepithelial connective tissue graft
  Arms: Test group: SCTG from tuberosity
Device: Intraoral optical scan — Intraoral optical scan was performed at both groups at baseline, 3 months, 4 months and 12 months to be able to compare volumetric changes.

SUMMARY:
The goal of this study is to compare clinical and histologically the soft tissue changes in terms of volume gain and stability around dental implants in cases where a subepithelial connective tissue graft from the palate or from the tuberosity is used randomly

DETAILED DESCRIPTION:
Understanding the importance of the soft tissue around implants have lead clinicians to develop surgical approaches to augment it. The majority of them, are described as bilaminar techniques obtaining a subephitelial connective tissue graft (SCTG) from the palate (P). However, recent studies have demonstrated that tuberosity (T) tissue is a very dense and coarse tissue that seems to contain more collagen and less fat and glandular tissue than that from the P, and therefore may have better tissue qualities for soft tissue augmentation, but there is limited scientific evidence comparing these areas.

The main goal of this study is to compare the soft tissue volume gain and stability around implants in cases where a SCTG of the same dimensions from the P or T is used randomly. To calculate volume changes and stability an intraoral optical scan is used and three-dimensional images superimposed.

The secondary goal is to compare histologically both tissues and changes in clinical parameters. Histomorphometry and immunohistochemistry evaluating levels of Type I-III collagen, long lysyl hydroxylase, matrix metalloproteinase 1-2, and monoclonal antibody against cytokeratin 4-10-13 is performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥18 years and able to understand the nature of the proposed surgery and to a signed informed consent.
* Implant must be located between 2 fixed reference points i.e. clinical crowns.
* All implants locations with a need of a soft tissue volume augmentation.
* Palate must have ≥2mm of thickness at premolar area.
* Tuberosity > 12mm in length.
* Full mouth plaque and bleeding score <20%.

Exclusion Criteria:

* Previous soft tissue augmentation in the area.
* Heavy Smokers (> 10 cigarettes per day).
* Local or systemic conditions that would interfere with routine periodontal therapy (non controlled diabetes, liver function disorder, immunosuppressant disease, autoimmune disease).
* Allergy to Non-Steroidal Anti-Inflammatory Drugs.
* Patients taking medications that cause gingival enlargement
* Gingival idiopatic overgrowth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Soft tissue volume gain | Baseline to 3 months postoperative
  Following soft tissue augmentation procedure volume gain is registered using intraoral optical scan. Superposition between three dimensional images from baseline (before augmentation procedure) and 3 months postoperative is done.
Soft tissue stability | 4 months postoperative to 12 months postoperative
  To evaluate soft tissue stability an intraoral optical scan is performed at 4 and 12 months postoperative. Also a superimposition between 4 months and 12 months optical images is done.

SECONDARY OUTCOMES:
Histology | Baseline
  Descriptive histology and immunohistochemistry evaluating: Type I-III collagen, long lysyl hydroxylase, matrix metalloproteinase 1-2, and monoclonal antibody against cytokeratin 4-10-13.
Clinical periodontal parameters Plaque Index and Bleeding on probing | Baseline, 3 months, 4 months, 12 months
  Plaque index, bleeding on probing expressed as a full mouth %.
Clinical periodontal parameters.Probing depth | Baseline, 3 months, 4 months, 12 months
  Probing depth expressed in mm. Evaluated at implant and adjacent teeth. At Mesial, distal, buccal, lingual, mesiobuccal, mesiolingual, distobuccal and distolingual levels.
Clinical periodontal parameters. Width of keratinized tissue | Baseline, 3 months, 4 months, 12 months
  Width of keratinized tissue expressed in mm, evaluated at medial point at implant and adjacent teeth one.

IPD SHARING:
Plan to Share IPD: No